CLINICAL TRIAL: NCT07010601
Title: U54 Pilot: Comparing Tobacco Product Susceptibility and Product Substitution by Relative Rurality and Alcohol Use
Brief Title: Tobacco Product Susceptibility and Substitutability by Rurality and Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark J Rzeszutek, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Mark J Rzeszutek, PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5U54DA058256-02 Pilot: #2345; 5U54DA058256-02 (NIH)
Record Dates: First submitted 2025-05-21; First posted 2025-06-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use; E-cigarette Use; Cigarette Use
MeSH Terms: conditions — Alcohol Drinking; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qualtrics and Experimental Tobacco Marketplace (Experimental): Participants who report using cigarettes/e-cigarettes will complete a Qualtrics survey consisting of various decision-making tasks, novel hypothetical nicotine product demand tasks, and Experimental Tobacco Marketplace scenarios (ETM). There will be three total ETM scenarios, cigarette adjusting price, e-cigarette adjusting price, and both e-cigarette and cigarette adjusting price.
  Interventions: Behavioral: Experimental Tobacco Marketplace; Behavioral: Hypothetical Novel Nicotine Product Purchase Tasks
- Qualtrics Only (Experimental): Participants who do not report using cigarettes/e-cigarettes will complete will complete a Qualtrics survey consisting of various decision-making tasks, and novel hypothetical nicotine product demand tasks
  Interventions: Behavioral: Hypothetical Novel Nicotine Product Purchase Tasks

INTERVENTIONS:
Behavioral: Experimental Tobacco Marketplace — This study will have three different scenarios in the Experimental Tobacco Marketplace (ETM) for participants who reported being cigarette and/or e-cigarette users. These will consist of hypothetical purchase scenarios where a variety of different tobacco products are available to purchase. The three ETM scenarios will be adjusting price cigarettes, adjusting price e-cigarettes, and both adjusting price cigarettes and e-cigarettes.
  Arms: Qualtrics and Experimental Tobacco Marketplace
Behavioral: Hypothetical Novel Nicotine Product Purchase Tasks — This study will have a set of hypothetical demand tasks for novel nicotine products. These tasks consist of different novel hypothetical products (combusted, oral, and vaporized) of differing nicotine content (high and low), and different flavors (preferred alcoholic flavor, no characterizing flavor) where likelihood to try is assessed at a variety of price points.

SUMMARY:
A high priority research area for the Food and Drug Administration Center for Tobacco Products (FDA CTP) is determining who will start using tobacco products and who will stop using tobacco products. A population that has a disproportionately high amount of tobacco use are people living in rural areas. This indicates that some aspect of rurality is related to tobacco product susceptibility and decreased tobacco cessation rates. People in rural areas also typically have higher rates of alcohol use, which is also associated with higher tobacco use and decreased tobacco cessation rates. The purpose of this study is to (1) examine how rurality and alcohol use may affect susceptibility to existing and novel tobacco products and (2) examine how rurality and alcohol use may affect likelihood for tobacco users to substitute to tobacco cessation products. To accomplish this, the investigators will use behavioral economic measures to assess how people respond to novel tobacco products (high and low nicotine, flavored and unflavored), as well as use the experimental tobacco marketplace to determine how current users might switch to products associated with cessation. Because rurality is a spectrum, the investigators will be using an index of relative rurality (IRR) to better quantify how rurality and alcohol use affect these tobacco-related behaviors.

ELIGIBILITY:
Cigarette/E-Cigarette Users

Inclusion Criteria:

* 21 years of age or older
* Smoke cigarettes or use e-cigarettes 25 or more days a month

Cigarette/E-Cigarette Non-Users

Inclusion Criteria:

* 21 years of age or older
* Do not report using an e-cigarette or cigarette in the past month

Risky Alcohol Users

Inclusion Criteria:

* 21 years of age or older
* A score of 8 or higher on the Alcohol Use Disorder Identification Test

Non-Risky Alcohol Users

Inclusion Criteria:

* 21 years of age or older
* A score of 7 or lower on the Alcohol Use Disorder Identification Test

All groups

Inclusion Criteria:

* Located in the USA
* At least 100 complete studies on Prolific

Exclusion Critera:

* Failing attention checks during the screener

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 737 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Demand Intensity and Price Sensitivity for Hypothetical Nicotine Products | Assessed at study week 0
  Likelihood to purchase and consume hypothetical nicotine products and sensitivity to cost of different product categories, flavors, and nicotine combinations will be assessed in all groups. Hypothetical demand will be assessed using non-linear mixed-effects modeling to obtain estimates of demand intensity and price sensitivity for these hypothetical products. Higher intensity and lower price sensitivity are indicators for higher subjective value and likelihood to try these novel products.
Alternative Product Purchasing as a Function of Change in Price of Cigarettes and/or E-Cigarettes in the Experimental Tobacco Marketplace | Assessed at study week 0
  Cigarette and e-cigarette users will complete different experimental tobacco marketplace scenarios. Alternative product purchasing (substitution) for different nicotine products as a function of increasing price of cigarettes/e-cigarettes will be measured with non-linear mixed-effects cross-commodity demand equations that determine the magnitude and direction of product substitution as a function of price increases of cigarettes and/or e-cigarettes. A higher magnitude indicates a larger change in product purchasing as a function of the ascending price item, where direction determines if the commodity was a complement to or substitute of the ascending price item(s). In the case of failures of non-linear model fitting, linear models will be used to determine product substitution based on intercept (initial purchasing) and slope (degree of substitution).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data from this study will be made as available as possible after acceptance for publication. All shared data will comply with HIPAA guidelines on personally identifiable information. Code used for analyses will also accompany deidentified data.
Supporting Information: Analytic Code

DOCUMENTS (1):
  • Informed Consent Form (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT07010601/ICF_000.pdf